CLINICAL TRIAL: NCT04373460
Title: Comparison of the Efficacy and Safety of Human Coronavirus Immune Plasma (HCIP) vs. Control (SARS-CoV-2 Non-immune) Plasma Among Outpatients With Symptomatic COVID-19
Brief Title: Convalescent Plasma to Limit SARS-CoV-2 Associated Complications
Acronym: CSSC-004
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: State of Maryland (Other Government); Bloomberg Philanthropies (Other); United States Department of Defense (U.S. Federal Agency); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00247590; R01AI152078 (NIH); W911QY2090012 (Other Grant/Funding Number: Department of Defense); U24TR001609 (NIH); UL1TR003098 (NIH)
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-01

CONDITIONS: SARS-CoV 2
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: A total of approximately 1344 eligible subjects stratified with a target goal (but not binding) of 50:50 in the <65 vs ≥ 65 age range will be randomized in a 1:1 ratio to receive either HCIP or control plasma.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SARS-CoV-2 convalescent plasma (Experimental): SARS-CoV-2 convalescent plasma (1 cup; minimum of 175 mL collected by apheresis from a volunteer who recovered from COVID-19 disease and has SARS-CoV-2 antibody titers ≥ 1:320 and after July 2021 meets FDA criteria for high titer plasma.
  Interventions: Biological: SARS-CoV-2 convalescent plasma
- Standard Control plasma (Active Comparator): Plasma collected from a volunteer donor prior to January 1, 2020 will not be tested for SARS-CoV-2 antibodies. Plasma collected after December 31, 2019 will be confirmed as SARS-CoV-2 seronegative.
  Interventions: Biological: Plasma from a volunteer donor

INTERVENTIONS:
Biological: SARS-CoV-2 convalescent plasma — SARS-CoV-2 convalescent plasma (1 cup; minimum of 175 mL collected by apheresis from a volunteer who recovered from COVID-19 disease and has SARS-CoV-2 antibody titers ≥ 1:320 and after July 2021 meets FDA criteria for high titer plasma.
  Other Names: Human coronavirus immune plasma (HCIP)
  Arms: SARS-CoV-2 convalescent plasma
Biological: Plasma from a volunteer donor — Plasma collected from a volunteer donor prior to January 1, 2020 will not be tested for SARS-CoV-2 antibodies. Plasma collected after December 31, 2019 will be confirmed as SARS-CoV-2 seronegative.
  Arms: Standard Control plasma

SUMMARY:
To assess the efficacy and safety of Human coronavirus immune plasma (HCIP) to reduce the risk of hospitalization or death, the duration of symptoms and duration of nasopharyngeal or oropharyngeal viral shedding.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blind, controlled, phase 2 trial is to evaluate the efficacy of treatment with HCIP in reducing hospitalization and death prior to hospitalization among outpatient adults who have RNA detection test-confirmed COVID-19 AND have developed any symptoms of COVID-19 including but not limited to fever, cough, or other COVID associated symptoms like anosmia. Ambulatory/outpatient adults subjects 18 years of age or older, regardless of risk factors for severe illness may participate. A total of approximately 1344 eligible subjects stratified with a target goal (but not binding) of 50:50 in the <65 vs ≥ 65 age range will be randomized in a 1:1 ratio to receive either HCIP or control plasma.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Competent and capable to provide informed consent
* • Positive molecular test for presence of SARS-CoV-2 in fluid collected by saliva for antigen, oropharyngeal or nasopharyngeal swab
* Experiencing any symptoms of COVID-19 including but not limited to fever(T> 100.5º F), cough, or other COVID associated symptoms like anosmia
* ≤ 8 days since the first symptoms of COVID-19
* ≤ 8 days since first positive SARS-CoV-2 RNA test
* Able and willing to comply with protocol requirements listed in the informed consent

Exclusion Criteria:

* Hospitalized or expected to be hospitalized within 24 hours of enrollment
* Psychiatric or cognitive illness or recreational drug/alcohol use that in the opinion of the principal investigator, would affect subject safety and/or compliance
* History of prior reactions to transfusion blood products
* Inability to complete therapy with the study product within 24 hours after enrollment
* Receiving any treatment drug for COVID-19 within 14 days prior to screening evaluation (monoclonal antibodies, compassionate use or study trial related). Steroid treatment at any time does not affect study eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1225 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Sullivan, MD, Principal Investigator — The Johns Hopkins University
Locations (29):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Center for American Indian Health - Chinle Office, Chinle, Arizona
  - Mayo Clinic, Phoenix, Phoenix, Arizona
  - University of Arizona, Phoenix, Tucson, Arizona
  - University of Arizona, Tuscon, Tucson, Arizona
  - Center for American Indian Health - Whiteriver Office, Whiteriver, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Irvine Health, Orange, California
  - Western Connecticut Health Network, Danbury Hospital, Danbury, Connecticut
  - Western Connecticut Health Network, Norwalk Hospital, Norwalk, Connecticut
  - University of Miami, Coral Gables, Florida
  - University of Miami Clinical Translational Research Site, Miami, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
  - Tulane University, New Orleans, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - The Johns Hopkins University, Baltimore, Maryland
  - MedStar Washington Hospital Center, Hyattsville, Maryland
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Center for American Indian Health - Gallup Office, Gallup, New Mexico
  - Center for American Indian Health - Shiprock Office, Shiprock, New Mexico
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Lifespan/BrownUniversity (Rhode Island Hospital), Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - The University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) collected in this study, including data dictionaries, will be made available to other researchers after the end of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of initial study manuscript
Access Criteria: Public

REFERENCES:
- [Result] Sullivan DJ, Gebo KA, Shoham S, Bloch EM, Lau B, Shenoy AG, Mosnaim GS, Gniadek TJ, Fukuta Y, Patel B, Heath SL, Levine AC, Meisenberg BR, Spivak ES, Anjan S, Huaman MA, Blair JE, Currier JS, Paxton JH, Gerber JM, Petrini JR, Broderick PB, Rausch W, Cordisco ME, Hammel J, Greenblatt B, Cluzet VC, Cruser D, Oei K, Abinante M, Hammitt LL, Sutcliffe CG, Forthal DN, Zand MS, Cachay ER, Raval JS, Kassaye SG, Foster EC, Roth M, Marshall CE, Yarava A, Lane K, McBee NA, Gawad AL, Karlen N, Singh A, Ford DE, Jabs DA, Appel LJ, Shade DM, Ehrhardt S, Baksh SN, Laeyendecker O, Pekosz A, Klein SL, Casadevall A, Tobian AAR, Hanley DF. Randomized Controlled Trial of Early Outpatient COVID-19 Treatment with High-Titer Convalescent Plasma. medRxiv [Preprint]. 2021 Dec 21:2021.12.10.21267485. doi: 10.1101/2021.12.10.21267485. PMID 34981068
- [Derived] Park HS, Yin A, Barranta C, Lee JS, Caputo CA, Sachithanandham J, Li M, Yoon S, Sitaras I, Jedlicka A, Eby Y, Ram M, Fernandez RE, Baker OR, Shenoy AG, Mosnaim GS, Fukuta Y, Patel B, Heath SL, Levine AC, Meisenberg BR, Spivak ES, Anjan S, Huaman MA, Blair JE, Currier JS, Paxton JH, Gerber JM, Petrini JR, Broderick PB, Rausch W, Cordisco ME, Hammel J, Greenblatt B, Cluzet VC, Cruser D, Oei K, Abinante M, Hammitt LL, Sutcliffe CG, Forthal DN, Zand MS, Cachay ER, Raval JS, Kassaye SG, Marshall CE, Yarava A, Lane K, McBee NA, Gawad AL, Karlen N, Singh A, Ford DE, Jabs DA, Appel LJ, Shade DM, Lau B, Ehrhardt S, Baksh SN, Shapiro JR, Ou J, Na YB, Knoll MD, Ornelas-Gatdula E, Arroyo-Curras N, Gniadek TJ, Caturegli P, Wu J, Ndahiro N, Betenbaugh MJ, Ziman A, Hanley DF, Casadevall A, Shoham S, Bloch EM, Gebo KA, Tobian AA, Laeyendecker O, Pekosz A, Klein SL, Sullivan DJ. Outpatient COVID-19 convalescent plasma recipient antibody thresholds correlated to reduced hospitalizations within a randomized trial. JCI Insight. 2024 Mar 14;9(8):e178460. doi: 10.1172/jci.insight.178460. PMID 38483534
- [Derived] Park HS, Yin A, Barranta C, Lee JS, Caputo CA, Sachithanandham J, Li M, Yoon S, Sitaras I, Jedlicka A, Eby Y, Ram M, Fernandez RE, Baker OR, Shenoy AG, Mosnaim GS, Fukuta Y, Patel B, Heath SL, Levine AC, Meisenberg BR, Spivak ES, Anjan S, Huaman MA, Blair JE, Currier JS, Paxton JH, Gerber JM, Petrini JR, Broderick PB, Rausch W, Cordisco ME, Hammel J, Greenblatt B, Cluzet VC, Cruser D, Oei K, Abinante M, Hammitt LL, Sutcliffe CG, Forthal DN, Zand MS, Cachay ER, Raval JS, Kassaye SG, Marshall CE, Yarava A, Lane K, McBee NA, Gawad AL, Karlen N, Singh A, Ford DE, Jabs DA, Appel LJ, Shade DM, Lau B, Ehrhardt S, Baksh SN, Shapiro JR, Ou J, Na YB, Knoll MD, Ornelas-Gatdula E, Arroyo-Curras N, Gniadek TJ, Caturegli P, Wu J, Ndahiro N, Betenbaugh MJ, Ziman A, Hanley DF, Casadevall A, Shoham S, Bloch EM, Gebo KA, Tobian AAR, Laeyendecker O, Pekosz A, Klein SL, Sullivan DJ. Outpatient COVID-19 convalescent plasma recipient antibody thresholds correlated to reduced hospitalizations within a randomized trial. medRxiv [Preprint]. 2023 Dec 15:2023.04.13.23288353. doi: 10.1101/2023.04.13.23288353. PMID 37131659
- [Derived] Baksh SN, Heath SL, Fukuta Y, Shade D, Meisenberg B, Bloch EM, Tobian AAR, Spivak ES, Patel B, Gerber J, Raval JS, Forthal D, Paxton J, Mosnaim G, Anjan S, Blair J, Cachay E, Currier J, Das P, Huaman M, Sutcliffe C, Yarava A, Casadevall A, Sullivan D, Hanley D, Gebo KA. Symptom Duration and Resolution With Early Outpatient Treatment of Convalescent Plasma for Coronavirus Disease 2019: A Randomized Trial. J Infect Dis. 2023 May 29;227(11):1266-1273. doi: 10.1093/infdis/jiad023. PMID 36722044
- [Derived] Sullivan DJ, Gebo KA, Shoham S, Bloch EM, Lau B, Shenoy AG, Mosnaim GS, Gniadek TJ, Fukuta Y, Patel B, Heath SL, Levine AC, Meisenberg BR, Spivak ES, Anjan S, Huaman MA, Blair JE, Currier JS, Paxton JH, Gerber JM, Petrini JR, Broderick PB, Rausch W, Cordisco ME, Hammel J, Greenblatt B, Cluzet VC, Cruser D, Oei K, Abinante M, Hammitt LL, Sutcliffe CG, Forthal DN, Zand MS, Cachay ER, Raval JS, Kassaye SG, Foster EC, Roth M, Marshall CE, Yarava A, Lane K, McBee NA, Gawad AL, Karlen N, Singh A, Ford DE, Jabs DA, Appel LJ, Shade DM, Ehrhardt S, Baksh SN, Laeyendecker O, Pekosz A, Klein SL, Casadevall A, Tobian AAR, Hanley DF. Early Outpatient Treatment for Covid-19 with Convalescent Plasma. N Engl J Med. 2022 May 5;386(18):1700-1711. doi: 10.1056/NEJMoa2119657. Epub 2022 Mar 30. PMID 35353960

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
Started | 610 | 615
Completed | 592 | 589
Not Completed | 18 | 26
Not completed — Did not receive tranfusion | 18 | 26

BASELINE CHARACTERISTICS:
Population: Includes participants who were randomized and received transfusion
Groups:
- Total: Total of all reporting groups
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma | Total
Number analyzed (Participants) | 592 | 589 | 1181
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [32 to 54] | 44 [33 to 55] | 43 [32 to 54]
Age, Customized [Count of Participants; unit: Participants]
  18 - 34 years | 190 | 165 | 355
  35 - 49 years | 207 | 208 | 415
  50 - 64 years | 155 | 176 | 331
  >=65 years | 40 | 40 | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 323 | 352 | 675
  Male | 269 | 237 | 506
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 80 | 90 | 170
  Not Hispanic or Latino | 512 | 499 | 1011
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 9 | 17
  Asian | 22 | 22 | 44
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 92 | 71 | 163
  White | 459 | 475 | 934
  More than one race | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
BMI category 1 [Count of Participants; unit: Participants]
  <30 | 382 | 355 | 737
  >=30 | 210 | 234 | 444
BMI category 2 [Count of Participants; unit: Participants]
  <35 | 495 | 482 | 977
  >=35 | 97 | 107 | 204
Hypertension [Count of Participants; unit: Participants]
  Yes | 140 | 136 | 276
  No | 452 | 453 | 905
Diabetes [Count of Participants; unit: Participants]
  Yes | 49 | 50 | 99
  No | 543 | 539 | 1082
Asthma [Count of Participants; unit: Participants]
  Yes | 59 | 73 | 132
  No | 533 | 516 | 1049
HIV infection [Count of Participants; unit: Participants]
  Yes | 13 | 12 | 25
  No | 579 | 577 | 1156
Pregnant [Count of Participants; unit: Participants]
  Yes | 2 | 1 | 3
  No | 590 | 588 | 1178
Time from symptom onset to transfusion [Median (Inter-Quartile Range); unit: days] | 6 [4 to 7] | 6 [4 to 7] | 6 [4 to 7]
Vaccine status [Count of Participants; unit: Participants]
  Unvaccinated | 486 | 479 | 965
  Partially vaccinated | 27 | 31 | 58
  Fully vaccinated | 79 | 79 | 158

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of Hospitalizations or Deaths Prior to Hospitalization
Description: Cumulative Number measured as the proportion of subjects who were hospitalized or who died prior to hospitalization
Time Frame: Up to day 28
Population: Includes patients who were randomized and received transfusion
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
Number analyzed (Participants) | 592 | 589
Participants | 17 | 37
Statistical Analysis 1: Comparison: SARS-CoV-2 Convalescent Plasma vs Standard Control Plasma; Test type: Superiority; p = 0.005, Fisher Exact; Risk Difference (RD) = 3.4, 95% CI 2-sided [1.0 to 5.8]

2. Primary Outcome: Cumulative Incidence of Severe Infusion Reactions
Description: Cumulative incidence measured as rate per person-years experiencing treatment-related severe infusion reactions during the study period.
Time Frame: Up to day 28
Population: Includes patients who were randomized and received transfusion
Measure: Number; unit: Rate per person-years
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
Number analyzed (Participants) | 592 | 589
Rate per person-years | 0.05 | 0.00
Statistical Analysis 1: Comparison: SARS-CoV-2 Convalescent Plasma vs Standard Control Plasma; Test type: Superiority; p = 0.16, Rate per person-years; Risk Difference (RD) = -0.05, 95% CI 2-sided [-0.11 to 0.02]

3. Primary Outcome: Cumulative Incidence of Treatment-related Grade 3 or Higher Adverse Events
Description: Cumulative incidence measured as rate per person-years experiencing a Grade 3 or higher.
Time Frame: Up to day 90
Measure: Number; unit: Rate per person-years
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
Number analyzed (Participants) | 592 | 589
Rate per person-years | 0.25 | 0.43
Statistical Analysis 1: Comparison: SARS-CoV-2 Convalescent Plasma vs Standard Control Plasma; Test type: Superiority; p = 0.02, Rate per person-years; Incidence rate difference = 0.18, 95% CI 2-sided [0.03 to 0.32]

4. Primary Outcome: Cumulative Incidence of Treatment-related Acute Respiratory Distress Syndrome (ARDS)
Description: Cumulative incidence measured as rate per person-years of treatment-related severe Acute Respiratory Distress Syndrome (ARDS) during the study period.
Time Frame: Up to day 28
Population: Includes patients who were randomized and received transfusion
Measure: Number; unit: Rate per person-years
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
Number analyzed (Participants) | 592 | 589
Rate per person-years | 0.00 | 0.01
Statistical Analysis 1: Comparison: SARS-CoV-2 Convalescent Plasma vs Standard Control Plasma; Test type: Superiority; p = 0.32, Rate per person-years; Risk Difference (RD) = 0.01, 95% CI 2-sided [-0.01 to 0.02]

5. Secondary Outcome: Serum SARS-CoV-2 Antibody Titers by Visit
Description: Geometric mean Spike Receptor Binding Domain (RBD) titers at day 0, 14, 28 and 90 between the randomized arms.
Time Frame: Days 0, 14, 28 and 90
Population: Analysis limited to those that were transfused and had the titer data performed
Measure: Geometric Mean (95% Confidence Interval); unit: Spike Receptor Binding Domain Titer
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
Number analyzed (Participants) | 577 | 564
Spike Receptor Binding Domain Titer
  Pre-transfusion | 345 [276 to 431] | 316 [254 to 393]
  Day 14: number analyzed (Participants) | 553 | 546
  Day 14 | 8595 [7211 to 10245] | 9868 [8217 to 11851]
  Day 28: number analyzed (Participants) | 541 | 534
  Day 28 | 10980 [9196 to 13111] | 12241 [10215 to 14668]
  Day 90: number analyzed (Participants) | 529 | 518
  Day 90 | 13958 [11577 to 16829] | 13281 [10979 to 16065]

6. Other Pre Specified Outcome: Number of Participants With ICU Admission
Description: Disease severity measured by admission to the ICU
Time Frame: Up to day 90
Population: Includes patients who were randomized and received transfusion
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
Number analyzed (Participants) | 592 | 589
Participants
  Admission to ICU | 3 | 7
  No admission to ICU | 589 | 582

7. Other Pre Specified Outcome: Number of Participants With Invasive Mechanical Ventilation
Description: Disease severity measured by invasive mechanical ventilation
Time Frame: Up to day 90
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
Number analyzed (Participants) | 592 | 589
Participants
  On invasive mechanical ventilation | 0 | 3
  No invasive mechanical ventilation | 592 | 586

8. Other Pre Specified Outcome: Number of Participants Who Died
Description: Disease severity measured by death
Time Frame: Up to day 90
Population: Includes patients who were randomized and received transfusion
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
Number analyzed (Participants) | 592 | 589
Participants
  Deaths | 0 | 3
  No deaths | 592 | 586

9. Other Pre Specified Outcome: Number of Participants With Resolved COVID-19 Symptoms at Day 14
Description: Number of participants with resolved COVID-19 symptoms at day 14
Time Frame: Day 14
Population: All participants who were transfused and had symptom data for day 14
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
Number analyzed (Participants) | 560 | 554
Participants | 146 | 134
Statistical Analysis 1: Comparison: SARS-CoV-2 Convalescent Plasma vs Standard Control Plasma; Test type: Superiority; p = 0.65, Fisher Exact

10. Other Pre Specified Outcome: Number of Participants With Resolved COVID-19 Symptoms at Day 28
Description: Number of participants with resolved COVID-19 symptoms at day 28
Time Frame: Day 28
Population: All participants who were transfused and had symptom data for day 28
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
Number analyzed (Participants) | 553 | 544
Participants | 250 | 245

11. Other Pre Specified Outcome: Number of Participants With Resolved COVID-19 Symptoms at Day 90
Description: Number of participants with resolved COVID-19 symptoms at day 90
Time Frame: Day 90
Population: All participants who were transfused and had symptom data for day 90
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
Number analyzed (Participants) | 533 | 528
Participants | 359 | 347

12. Other Pre Specified Outcome: Impact of Convalescent Plasma on Outcome as Assessed by Change in Hospitalization Rate
Description: Assess change in hospitalization rate as measured by number of hospitalizations stratified by age groups <65 and >=65
Time Frame: Day 0 to Day 90
Population: Includes patients who were randomized and received transfusion
Measure: Count of Participants; unit: Participants
Groups:
- SARS-CoV-2 Convalescent Plasma Total Age < 65: SARS-CoV-2 convalescent plasma (1 cup; minimum of 175 mL collected by apheresis from a volunteer who recovered from COVID-19 disease and has SARS-CoV-2 antibody titers ≥ 1:320 and after July 2021 meets FDA criteria for high titer plasma.
  SARS-CoV-2 convalescent plasma: SARS-CoV-2 convalescent plasma (1 cup; minimum of 175 mL collected by apheresis from a volunteer who recovered from COVID-19 disease and has SARS-CoV-2 antibody titers ≥ 1:320 and after July 2021 meets FDA criteria for high titer plasma.
- Standard Control Plasma Total Age <65: Plasma collected from a volunteer donor prior to January 1, 2020 will not be tested for SARS-CoV-2 antibodies. Plasma collected after December 31, 2019 will be confirmed as SARS-CoV-2 seronegative.
  Plasma from a volunteer donor: Plasma collected from a volunteer donor prior to January 1, 2020 will not be tested for SARS-CoV-2 antibodies. Plasma collected after December 31, 2019 will be confirmed as SARS-CoV-2 seronegative.
Arm/Group | SARS-CoV-2 Convalescent Plasma Total Age < 65 | Standard Control Plasma Total Age <65
Number analyzed (Participants) | 592 | 589
Participants
  Age group < 65: number analyzed (Participants) | 552 | 549
  Age group < 65: Primary event of hospitalization | 12 | 29
  Age group < 65: No primary event of hospitalization | 540 | 520
  Age group >= 65: number analyzed (Participants) | 40 | 40
  Age group >= 65: Primary event of hospitalization | 5 | 8
  Age group >= 65: No primary event of hospitalization | 35 | 32

13. Other Pre Specified Outcome: Impact of Donor Antibody Titers on Hospitalization Rate of Convalescent Plasma Recipients
Description: Impact of donor antibody titers (high/low) will be assessed by hospitalization rate as measured by number of hospitalizations.
Time Frame: Day 0 to Day28
Population: Analysis limited to those that had the donor titer measured
Measure: Count of Participants; unit: Participants
Groups:
- SARS-CoV-2 Convalescent Plasma (High Titer): High titer refers >= median donor dilutional neutralizing virus titer
- SARS-CoV-2 Convalescent Plasma (Low Titer): Low titer refers to < median donor dilutional neutralizing virus titer
Arm/Group | SARS-CoV-2 Convalescent Plasma (High Titer) | SARS-CoV-2 Convalescent Plasma (Low Titer)
Number analyzed (Participants) | 302 | 264
Participants
  Hospitalized | 6 | 10
  Not hospitalized | 296 | 254
Statistical Analysis 1: Comparison: SARS-CoV-2 Convalescent Plasma (High Titer) vs SARS-CoV-2 Convalescent Plasma (Low Titer); Test type: Superiority; Risk Ratio (RR) = 0.525, 95% CI 2-sided [0.192 to 1.425]

ADVERSE EVENTS:
Time Frame: 90 days
Description: We have analyzed adverse event on the severity grade system 1 through 5, with grades 3-5 categorized as severe.
Arm/Group | SARS-CoV-2 Convalescent Plasma | Standard Control Plasma
All-Cause Mortality (participants affected / at risk) | 0/592 | 3/589
Serious Adverse Events (participants affected / at risk) | 34/592 | 55/589
Other Adverse Events (participants affected / at risk) | 106/592 | 109/589
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SARS-CoV-2 Convalescent Plasma (N=592) | Standard Control Plasma (N=589)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Kidney Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 14 (14) | 31 (31)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 4 (4) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SARS-CoV-2 Convalescent Plasma (N=592) | Standard Control Plasma (N=589)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 1 (1)
Burning and itching eyes (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Left Lower Eyelid Edema (Eye disorders) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 2 (2)
Fever (General disorders) | 3 (3) | 2 (2)
Heavy chest pain feeling (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 2 (2)
Pain (General disorders) | 2 (2) | 0 (0)
Worsening Anxiety (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2)
Post-vaccine reaction (Immune system disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Shingles (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 4 (4)
Vaginal infection (Infections and infestations) | 2 (2) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Facial contusions secondary to assault (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 13 (13) | 15 (15)
Laceration of Forehead (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Alcohol intolerance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms in lower extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Right knee sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Twitch in lip (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Renal calculi (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 9 (9) | 10 (10)
Hypertension (Vascular disorders) | 4 (4) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT04373460/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT04373460/SAP_001.pdf
  • Informed Consent Form (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT04373460/ICF_002.pdf